CLINICAL TRIAL: NCT01469546
Title: Phase II Trial Evaluating Axitinib (AG-013736) In Patients With Unresectable, Recurrent Or Metastatic Head And Neck Cancer
Brief Title: Phase II Trial Evaluating Axitinib In Patients With Unresectable, Recurrent Or Metastatic Head And Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2011.053; HUM00051095 (Other: University of Michigan IRB Number)
Record Dates: First submitted 2011-10-24; First posted 2011-11-10 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axitinib (AG-013736) (Experimental): A prospective, single-institution, single-arm phase II study of Axitinib in patients with unresectable recurrent and metastatic head and neck squamous cell carcinoma who have received no more than two prior lines of systemic therapy for recurrent or metastatic head and neck cancer.
  Interventions: Drug: Axitinib (AG-013736)

INTERVENTIONS:
Drug: Axitinib (AG-013736) — The subjects will be started on treatment with 5 mg of Axitinib twice a day continuously, with subsequent dose escalation to 7 mg and then 10 mg twice a day in the absence of grade 2 or worse toxicities. This will be followed by clinical and/or radiologic response assessment after 8 weeks and subsequently every 2 months until disease progression (defined per RECIST [Response Evaluation Criteria In Solid Tumors] criteria, or obvious progression on clinical or laryngoscopic/endoscopic exam) or intolerable toxicity (defined as below). During treatment on this protocol, all patients will be evaluated for safety. Correlative biomarker analysis will also be conducted.

SUMMARY:
The purpose of this study is to investigate a new agent Axitinib in the treatment of head and neck cancer.

This is a new drug that is given as a pill twice a day to treat cancer. This is one of the new, "smart" drugs. It binds to a protein on the surface of the cancer cell called VEGFR, and this way it slows down the growth of cancer cells and kills them. Head and neck cancer cells are known to carry this protein on their surface. Research in animals and in patients with other kinds of cancer showed that Axitinib can be effective at killing cancer cells, or stopping their growth, by this mechanism. It is generally a safe drug that is given by mouth. The investigators do not know, however, whether Axitinib is effective in head and neck cancer. This research study is being conducted to learn if Axitinib works in head and neck cancer, and also to learn to predict who would benefit from it. Four blood draws will be done to check special blood tests while the subjects are treated with Axitinib. These will be drawn at the same time as your routine labs, and there will not be additional sticks needed. A biopsy of the tumor before and after 1 month of treatment may be obtained to test how the cancer cells are responding to treatment. By testing these blood and tissue samples, the researchers will look at special tests (protein molecules) to try to determine what kind of head and neck patients would best respond to this drug. This is an open-label study, meaning that all subjects are on the active drug and there is no placebo (sugar pill).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically documented squamous cell head and neck cancer with or without metastases, not amenable to curative treatment.
2. Presence of measurable disease by CT scan.
3. Adequate bone marrow, hepatic, and renal function (including absence of proteinuria, PT (Prothrombin Time) <1.5, WBC (White Blood Cell count)≥ 3x109 cells/ml, ANC (Absolute Neutrophil Count) ≥ 1.5x109 cell/ml, platelets ≥75,000 cells/mm3, hemoglobin ≥ 9.0 g/dL, concentrations of total serum bilirubin within 1.5 x upper limit of normal (ULN), AST (Aspartate Aminotransferase), ALT (Alanine Aminotransferase) within 2.5x institutional upper limits of normal unless there are liver metastases in which case AST and ALT within 5.0 x ULN, serum creatinin clearance ≥ 60 ml/min), urinary protein <2+ by urine dipstick (if dipstick is ≥2+ then a 24-hour urine collection can be done and the patient may enter only if urinary protein is <2 g per 24 hours), documented within 14 days prior to initiation of Axitinib treatment.
4. Age ≥18 years.
5. ECOG (Eastern Cooperative Oncology Group) performance status of 0-2.
6. Life expectancy of ≥12 weeks.
7. No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 30 minutes apart. The baseline systolic blood pressure readings must be ≤140 mm Hg, and the baseline diastolic blood pressure readings must be ≤90 mm Hg. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
8. Women of childbearing potential must have a negative serum or urine pregnancy test within 3 days prior to treatment.
9. Signed and dated informed consent document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment.
10. Willingness and ability to comply with scheduled visits, treatment plans, including willingness to take Axitinib, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Central lung lesions involving major blood vessels (arteries or veins) or a tumor encasing major blood vessels (i.e. carotid artery).
2. History of hemoptysis.
3. Gastrointestinal abnormalities causing impaired absorption requiring intravenous alimentation, prior surgical procedures affecting absorption including gastric resection, treatment for active peptic ulcer disease in the past 6 months, active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy, malabsorption syndromes.
4. Previous treatment with anti-angiogenesis agents including thalidomide, or inhibitors of epidermal growth factor (EGF), platelet derived growth factor (PDGF), or fibroblast growth factors (FGF) receptors within 30 days preceding study entrance.
5. Current use or anticipated inability to avoid use of drugs that are known potent CYP3A4 inhibitors (ie, grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, clarithromycin, telithromycin, ergot derivatives, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, atazanavir, amprenavir, fosamprenavir , and delavirdine).
6. Current use or anticipated inability to avoid use of drugs that are known CYP3A4 or CYP1A2 inducers (ie, carbamazepine, felbamate, omeprazole, phenobarbital, phenytoin, amobarbital, nevirapine, primidone, rifabutin, rifampin, and St. John's wort).
7. Active seizure disorder or evidence of brain metastases, spinal cord compression, or carcinomatous meningitis.
8. A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment.
9. History of a malignancy (other than head and neck cancer) except those treated with curative intent for skin cancer (other than melanoma), in situ breast or in situ cervical cancer, or those treated with curative intent for any other cancer with no evidence of disease for 2 years.
10. Major surgery <4 weeks or radiation therapy <2 weeks of starting the study treatment. Prior palliative radiotherapy to metastatic lesion(s) is permitted, provided there is at least one measurable lesion that has not been irradiated.
11. Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
12. Patients (male and female) having procreative potential who are not willing or not able to use adequate contraception or practicing abstinence.
13. Women who are pregnant or breast-feeding.
14. History of prior treatment with more than 2 lines of therapy for metastatic head and neck cancer.
15. Patients with history of bleeding diathesis, DVT (deep venous thrombosis) or arterial thromboembolism, current use of therapeutic anticoagulation with oral vitamin K antagonists, factor Xa inhibitors, heparin products, oral direct thrombin inhibitors, or presence of non-healing wounds. Low-dose anticoagulants for maintenance of patency of central venous access device or prevention of deep venous thrombosis is allowed.
16. Patients residing in prison.
17. Prior experimental therapy within 30 days of planned start of this trial.
18. HIV virus infection irrespective of viral load, treatment status, or CD4 count, or acquired immunodeficiency syndrome (AIDS)-related illness.
19. Any of the following within the 12 months prior to study drug administration: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack.
20. History of deep vein thrombosis or pulmonary embolism within 6 month of anticipated starting of Axitinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-01; Primary Completion 2015-04 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis P Worden, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 42 patients were enrolled. 12 patients did not complete the first cycle or undergo repeat tumor imaging (due to adverse event, disease progression, non-compliance or physician discretion). Only 30 patients were analyzed..
Groups:
- Axitinib (AG-013736): Axitinib (AG-013736): The subjects will be started on treatment with 5 mg of Axitinib twice a day continuously, with subsequent dose escalation to 7 mg and then 10 mg twice a day in the absence of grade 2 or worse toxicities.
Period: Received 5 mg Dose
Arm/Group | Axitinib (AG-013736)
Started | 42
Completed First Cycle | 30
Completed | 19
Not Completed | 23
Not completed — Adverse Event | 13
Not completed — Death | 2
Not completed — Protocol Violation | 2
Not completed — Progressive Disease | 3
Not completed — Physician Decision | 3
Period: Dose Escalation to 10 mg
Arm/Group | Axitinib (AG-013736)
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 42 patients were enrolled. 12 patients did not complete the first cycle or undergo repeat tumor imaging (due to adverse event, disease progression, non-compliance or physician discretion). Only 30 patients were analyzed.
Arm/Group | Axitinib (AG-013736)
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 62 [40.0 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Alive and Free of Progression at 6 Months
Description: To determine the 6-months progression-free survival (PFS) rate in patients with unresectable recurrent and metastatic head and neck cancer treated with Axitinib.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number; unit: percentage of patients
Arm/Group | Axitinib (AG-013736)
Number analyzed (Participants) | 30
percentage of patients | 27

2. Secondary Outcome: Number of Participants Who Achieved Complete Response, Partial Response or Stable Disease
Description: To determine the disease control rate (complete response+partial response+stable disease), in patients with unresectable recurrent and metastatic head and neck cancer treated with Axitinib.
  Response Evaluation Criteria in Solid Tumors (RECIST version 1.0) will be used.
  Complete Response is defined as the disappearance of all tumor for a period of one month.
  Partial Response is defined as a 30% or more decrease in the sum of the longest diameters (LD) of all measured lesions without any evidence of progression of any lesion or the appearance of any new lesion for a period of one month.
  Stable Disease is defined as any change in measurable disease which is less than the criteria for partial remission or progression without any evidence of new lesions and persisting for at least 2 evaluations or 2 months.
Time Frame: 2 years
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | Axitinib (AG-013736)
Number analyzed (Participants) | 30
participants | 23

3. Secondary Outcome: Number of Patients That Experienced Grade 3 or 4 Toxicities
Description: The number of patients who develop these while on treatment and for 28 days after cessation of axitinib, and graded in severity per CTCAE v. 3.0 and as described in the protocol. According to the CTCAE v. 3.0, grade 3 toxicities are severe and grade 4 toxicities are life-threatening or disabling.
Time Frame: 28 Days Post Treatment
Population: All patients that received at least one dose of treatment were analyzed for toxicity.
Measure: Number; unit: patients
Arm/Group | Axitinib (AG-013736)
Number analyzed (Participants) | 42
patients
  Fatigue | 7
  Rash | 5
  Mucocitis/Stomatitis | 3
  Pain | 1
  Thrombosis | 1

4. Secondary Outcome: Median Progression-Free Survival (PFS)Time
Description: To evaluate PFS time in patients with Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (R/M SCCHN) treated with Axitinib.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Axitinib (AG-013736)
Number analyzed (Participants) | 30
months | 3.7 [3.5 to 5.7]

ADVERSE EVENTS:
Description: All 42 patients received treatment and were therefore evaluable for adverse events.
Arm/Group | Axitinib (AG-013736)
Serious Adverse Events (participants affected / at risk) | 22/42
Other Adverse Events (participants affected / at risk) | 37/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib (AG-013736) (N=42)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Cardiac ischemia/infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Death not associated with CTCAE term (General disorders) | 6 (6)
Dehydration (Gastrointestinal disorders) | 1 (1)
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1 (1)
Obstruction, GI (Gastrointestinal disorders) | 1 (1)
Stricture/stenosis (including anastomotic), GI (Gastrointestinal disorders) | 1 (1)
Hemorrhage, GI (Vascular disorders) | 3 (3)
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 2 (2)
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 1 (1)
Infection, Lung (Infections and infestations) | 1 (1)
Infection, Blood (Infections and infestations) | 1 (1)
Infection, Skin (Infections and infestations) | 1 (1)
Infection with unknown ANC, Lung (Infections and infestations) | 2 (2)
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Pain, Abdomen (Gastrointestinal disorders) | 1 (1)
Pain, Chest (General disorders) | 2 (2)
Pain, Eye (Eye disorders) | 1 (2)
Pain, Face (General disorders) | 1 (1)
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axitinib (AG-013736) (N=42)
Allergic reaction/hypersensitivity (Immune system disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 7 (10)
Pericardial effusion (non-malignant) (Cardiac disorders) | 1 (1)
Constitutional Symptoms (General disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 26 (40)
Fever (in the absence of neutropenia) (General disorders) | 1 (1)
Weight loss (General disorders) | 9 (12)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (2)
Rash/desquamation (Immune system disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4 (12)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 8 (10)
Constipation (Gastrointestinal disorders) | 8 (10)
Dehydration (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 11 (16)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3 (3)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 4 (4)
Fistula, GI (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (3)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 2 (2)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 3 (3)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 11 (18)
Nausea (Gastrointestinal disorders) | 6 (6)
Vomiting (Gastrointestinal disorders) | 2 (2)
Hemorrhage, GI (Vascular disorders) | 1 (1)
Hemorrhage, GI (Vascular disorders) | 2 (3)
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 1 (1)
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 1 (2)
Infection - Other (Infections and infestations) | 2 (2)
Infection, Bronchus (Infections and infestations) | 1 (1)
Infection, Pneumonia (Infections and infestations) | 1 (1)
Infection, Paranasal (Infections and infestations) | 2 (3)
Infection, Upper Airway (Infections and infestations) | 1 (1)
Infection, Urinary Tract (Infections and infestations) | 1 (1)
Edema: head and neck (Blood and lymphatic system disorders) | 1 (2)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Proteinuria (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spine-range of motion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Mood alteration (Nervous system disorders) | 2 (2)
Neurology (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 1 (2)
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1)
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 1 (1)
Watery eye (epiphora, tearing) (Eye disorders) | 1 (1)
Pain, Abdomen (Gastrointestinal disorders) | 3 (3)
Pain, Back (Musculoskeletal and connective tissue disorders) | 3 (6)
Pain, Chest (General disorders) | 3 (4)
Pain, External Ear (Ear and labyrinth disorders) | 1 (1)
Pain, Head (Nervous system disorders) | 7 (9)
Pain, Muscle (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain, Neck (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain, Oral Cavity (Gastrointestinal disorders) | 10 (13)
Pain, NOS (General disorders) | 2 (2)
Pain, Throat (Gastrointestinal disorders) | 3 (5)
Pain - Other (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (2)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes